CLINICAL TRIAL: NCT03794505
Title: Health Related Quality of Life and Pain Managment Using Infiltration or Suprascapular Nerve Block Ultrasound Guided in Patients With Glenohumeral Arthirtis
Brief Title: Quality of Life and Pain With Infiltration or Suprascapular Nerve Block in Glenohumeral Arthirtis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Luis Alonso Calderon Cordova, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F-2018-3401-056
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Shoulder Arthritis
MeSH Terms: interventions — Methylprednisolone Acetate; Lidocaine; Ropivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder infiltration (Active Comparator): Shoulder infiltration using 2 ml of Lidocaine 2% Injectable Solution and methylprednisolone acetate 40 mg
  Interventions: Drug: Methylprednisolone Acetate; Drug: Lidocaine 2% Injectable Solution
- Suprascapular nerve block (Experimental): Suprascapular nerve block ultrasound guided using 25 mg of Ropivacaine HCl Inj 7.5 MG/ML and methylprednisolone acetate 40 mg
  Interventions: Drug: Methylprednisolone Acetate; Drug: Ropivacaine HCl Inj 7.5 MG/ML

INTERVENTIONS:
Drug: Methylprednisolone Acetate — depo-medrol 40 mg
  Other Names: depo-medrol 40 mg
Drug: Lidocaine 2% Injectable Solution — 2ml of 2% lidocaine
  Other Names: xilocaine
  Arms: Shoulder infiltration
Drug: Ropivacaine HCl Inj 7.5 MG/ML — 25 mg
  Other Names: Ropivacaine
  Arms: Suprascapular nerve block

SUMMARY:
Efficacy in pain and health related quality of life of suprascapular nerve block ultrasound guided and glenohumeral infiltration in glenohumeral arthritis

DETAILED DESCRIPTION:
To describe the efficacy in pain management and health related quality of life of suprascapular nerve block ultrasound guided and glenohumeral infiltration in patients with glenohumeral arthritis

ELIGIBILITY:
Inclusion Criteria:

* IMSS affiliated
* Glenohumeral arthritis diagnosed

Exclusion Criteria:

* Previusly treatment for the same disease
* No follow up
* Dead

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Pain before | VAS before intervention
  visual analogue scale
Pain 2 months after | VAS 2 months after
  Visual analogue scale 2 months after procedure
Pain 6 months after | VAS 6 months after
  Visual analogue scale 6 months after procedure

SECONDARY OUTCOMES:
Quality of life before procedure | SF12v2 before procedure
  SF12v2 Health related quality of life before procedure
Quality of life 2 months after procedure | SF12v2 2 months after
  SF12v2 Health related quality of life 2 months after
Quality of life 6 months after procedure | SF12v2 6 months after
  SF12v2 Health related quality of life 6 months after

CONTACTS AND LOCATIONS:
Overall Officials: Luis Alonso Calderon Cordova, MD, Principal Investigator — IMSS
Locations (1):
- Department of Orthopedics, UMAE "Dr. Victorio de la Fuente Narváez" IMSS-UNAM. Ciudad de México, México, Mexico City, Gustavo A Madero, Mexico

IPD SHARING:
Plan to Share IPD: No